CLINICAL TRIAL: NCT01981057
Title: Clinical Experience With Numeta- Impact on Intake of Nutrients and Costs
Brief Title: Clinical Experience With Numeta in Preterm Infants
Acronym: Numeta
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoc.Prof.MD, Medical University of Vienna
Other Study IDs: MUV-Numeta
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2014-05

CONDITIONS: Premature Infants
Keywords: parenteral nutrition; Numeta; prescription software Cato Pan
MeSH Terms: conditions — Premature Birth; Hyperphagia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Numeta: parenteral receipt prescribed with Numeta
  Interventions: Other: Numeta; Other: Individual
- Individual: individually prescribed parenteral receipt
  Interventions: Other: Numeta; Other: Individual

INTERVENTIONS:
Other: Numeta — parenteral receipt prescribed with Numeta
Other: Individual — parenteral receipt prescribed individually

SUMMARY:
The aim of this prospective noninterventional study is to evaluate the clinical application of Numeta® in preterm infants and critically ill neonates in comparison to individualized prescribed parenteral nutrition. With the prescription software Cato-PAN® (by Cato software solutions) exact valid prescriptions for ordering parenteral nutrition solutions for premature infants are compared. Each PN solution is prescribed individually as well as with Numeta. Prescriptions were mirrored with respect to weight, venous approach, total volume and amount of enteral feeding, 24h medication and flipped vice versa. The key nutrient for calculating Numeta prescriptions was protein. The results of PN prescriptions were compared with each other/ESPGHAN recommendations. The investigators hypothesize that nutrimental content of Numeta prescriptions is equal to individually prescribed .parenteral nutrition solutions

ELIGIBILITY:
Inclusion Criteria:

* preterm infants <37 weeks gestational age
* parenteral nutrition therapy

Exclusion Criteria:

* hypersensitivity to egg, soy or peanut proteins or to any of the active substances
* congenital abnormality of the amino acid metabolism
* pathogenically elevated plasma concentrations of sodium, potassium, magnesium, calcium and/or phosphorous
* severe hyperglycemia
* severe hyperlipidemia
* severe disorders of lipid metabolism characterized by hypertriglyceridemia

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kreissl A, Repa A, Binder C, Thanhaeuser M, Jilma B, Berger A, Haiden N. Clinical Experience With Numeta in Preterm Infants: Impact on Nutrient Intake and Costs. JPEN J Parenter Enteral Nutr. 2016 May;40(4):536-42. doi: 10.1177/0148607115569733. Epub 2015 Feb 5. PMID 25655621

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Numeta | Individual
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Numeta | Individual | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Full Range); unit: days of gestation] | 233 [189 to 283] | 233 [189 to 283] | 233 [189 to 283]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  Austria | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Protein
Description: Prescriptions for protein in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: g/kg/d
Arm/Group | Numeta | Individual
Number analyzed (Participants) | 50 | 50
g/kg/d | 3.1 [1.6 to 4.1] | 3.6 [1.7 to 5]

2. Secondary Outcome: Energy
Description: Prescriptions for energy in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Carbohydrates
Description: Prescriptions for carbohydrates in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Fat
Description: Prescriptions for fat in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Sodium
Description: Prescriptions for sodium in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Potassium
Description: Prescriptions for Potassium in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Calcium
Description: Prescriptions for calcium in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Magnesium
Description: Prescriptions for magnesium in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Phosphorous
Description: Prescriptions for phosphorous in parenteral nutrition solutions will be ordered individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Osmolarity
Description: Osmolarity in parenteral nutrition solutions will be calculated individually and flipped with Numeta or "vice versa". This mirroring will be performed with the Cato-Pan prescription software. Subsequently the following nutrients will be calculated and compared with each other and with the ESPGHAN recommendations
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Numeta | Individual
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes